CLINICAL TRIAL: NCT04070573
Title: A Randomized Controlled Trial Comparing Low Doses Of Aspirin In The Prevention Of Preeclampsia (ASAPP)
Brief Title: Low Doses of Aspirin in the Prevention of Preeclampsia
Acronym: ASAPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-05020160
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Preeclampsia
Keywords: Preterm preeclampsia; Preeclampsia with severe features; High risk pregnancy; Low dose aspirin; Cell free RNA; Compliance
MeSH Terms: conditions — Pre-Eclampsia; Patient Compliance | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Arm 1: 81mg oral ASA daily. Arm 2: 162mg oral ASA daily. Patients will obtain their prescriptions from their respective pharmacies. Women in Arm 1, will be instructed to take one table of 81mg aspirin per day; those in Arm 2, will be asked to take two tablets simultaneously orally once per day. Therapy will be initiated at the baseline visit and continued until 1 week before planned delivery or upon admission for unplanned/imminent delivery as per clinical routine.
Who Masked: Outcomes Assessor
Masking Description: This is an open label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 81mg ASA (Active Comparator): Patients in Arm 1, will be instructed to take one tablet of 81mg aspirin per day.
  Interventions: Drug: acetylsalicylic acid
- 162mg ASA (Active Comparator): Patients in Arm 2, will be instructed to take two tablets simultaneously orally once per day.
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: acetylsalicylic acid — High risk pregnant women will be treated with daily aspirin during pregnancy.
  Other Names: aspirin; ASA

SUMMARY:
Preeclampsia (PE) is a morbid and potentially lethal complication of pregnancy and is more common in women with specific risk factors. Aspirin (ASA) is currently the only prophylactic therapy for preeclampsia in high-risk women to be recognized by the US Preventive Task Force and should be initiated early in the second trimester of pregnancy, before 16 weeks of gestation. However, currently there is no literature comparing various low-dose ASA formulations in the risk reduction of PE. In the United States, the currently available low-dose ASA is over the counter and is found in 81mg tablets. Therefore, when clinicians initiate therapy with low dose ASA, they may prescribe 1 or 2 tablets of 81mg aspirin per day depending on personal preference and cannot be assisted by evidence to guide their decision.This study aims to determine the incidence of preterm PE or PE with severe features in women taking either 81mg or 162mg in a randomized setting, from a single center. The investigators hypothesize that the information gained from this trial will permit a more accurate sample size calculation for a larger clinical trial powered to accept or reject our testing hypothesis. If our hypothesis is rejected and 162mg of daily ASA is not associated with a lower incidence of severe or preterm PE compared to 81mg, this may be due to lack of power to detect a smaller effect. The investigators would then evaluate the feasibility and results and determine whether a larger trial is reasonable.

DETAILED DESCRIPTION:
Preeclampsia (PE) is a serious and potentially fatal complication of pregnancy. It is a placental disease characterized by an elevated blood pressure in the 3rd trimester with multisystem involvement (proteinuria, elevated liver enzymes, low platelet count and/or neurologic symptoms). PE can cause pulmonary edema, seizures, or stroke and is a leading cause of maternal mortality. The pregnancy outcomes are further worsened if PE develops before term. Women who have a history of PE in a prior pregnancy, diabetes, preexisting hypertension, kidney disease, multifetal gestation or autoimmune diseases are at an increased risk to develop PE in a subsequent pregnancy.

Clinical trials evaluating the benefits of low-dose aspirin (ASA) have used a wide range of doses from 60mg to 150mg orally daily with low-dose being defined as less than 325mg per day. Taking ASA (as opposed to placebo) is thought to reduce the risk of preeclampsia by 17%, without increasing the risk of major obstetric bleeding. The number needed to treat is only 19 women. ASA is currently the only prophylactic therapy for PE in high-risk women to be recognized by the US Preventive Task Force and should be initiated early in the second trimester of pregnancy, before 16 weeks of gestation.

There has also been more awareness that the efficacy of ASA in preventing preeclampsia is limited by the poor adherence of patients to this therapy. Indeed, a cross-sectional study has estimated that up to 46% of women (n=42) on ASA therapy may not be compliant to it, as determined by a validated Simplified Medication Adherence Questionnaire (SMAQ). Adherence is essential to the efficacy of ASA in preventing preterm preeclampsia. It would therefore be of interest to obtain more information about adherence to ASA in women who need this therapy.

Assessing molecular pathways in the development of PE may allow opportunity for earlier diagnosis, specific triaging of patients to closer monitoring and further development of preventative or curative treatment strategies. Samples will be biobanked for biomarker discovery in the future.

The current literature is lacking in evidence to recommend a specific daily dose of ASA. Recent meta-analyses have suggested that there may be a dose response in the protective effect of ASA for PE. As compared to 60mg per day, an ASA dose of 100mg per day was associated with a lower relative risk of PE (0.44 vs 0.57, p=0.36). A large study of 1776 women has compared a slightly higher dose of ASA (150mg per day) to placebo and found a decrease in preterm delivery (before 37 weeks) due to PE (OR 0.38, p=0.004). Meta-analyses have shown that any dose of ASA above 60mg per day is protective and should be used to prevent PE in high risk pregnancies.

To date, there has not been any studies comparing lower doses of ASA (such as 81mg, the traditional "baby aspirin" dose sold in the US) to higher "low-dose" ASA regimens (such as 162mg) in their ability to prevent preterm or severe PE in women who are at a high risk for this devastating disease.

ELIGIBILITY:
Patients are currently only being enrolled at the New York Presbyterian Weill Cornell Medicine and at the New York Presbyterian Queens campuses.

Inclusion Criteria:

Pregnant patients, ≥18 years old, at less than 16 weeks' gestation (as documented by ultrasound) with at least one of the following risk factors for developing PE:

* PE in a prior pregnancy
* Chronic hypertension (prior to pregnancy or before 20 weeks' gestation)
* Type 1 or 2 diabetes
* Renal disease (proteinuria ≥300mg/day or estimated GFR<90mL/min/1.73 m2)
* Multifetal gestation
* Autoimmune disease (e.g. systemic lupus erythematous, antiphospholipid syndrome)

Exclusion Criteria:

* Patient with known intention to terminate pregnancy
* Major fetal malformation seen on ultrasound
* Contraindication to ASA therapy (including but not limited to allergy and high bleeding risk)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Line Malha, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York Presbyterian - Weill Cornell, New York, New York
  - New York Presbyterian Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Lisonkova S, Joseph KS. Incidence of preeclampsia: risk factors and outcomes associated with early- versus late-onset disease. Am J Obstet Gynecol. 2013 Dec;209(6):544.e1-544.e12. doi: 10.1016/j.ajog.2013.08.019. Epub 2013 Aug 22. PMID 23973398
- [Background] Duley L, Henderson-Smart DJ, Meher S, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004659. doi: 10.1002/14651858.CD004659.pub2. PMID 17443552
- [Background] Henderson JT, Whitlock EP, O'Conner E, Senger CA, Thompson JH, Rowland MG. Low-Dose Aspirin for the Prevention of Morbidity and Mortality From Preeclampsia: A Systematic Evidence Review for the U.S. Preventive Services Task Force [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Apr. Report No.: 14-05207-EF-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK196392/ PMID 24783270
- [Background] Abheiden CN, van Reuler AV, Fuijkschot WW, de Vries JI, Thijs A, de Boer MA. Aspirin adherence during high-risk pregnancies, a questionnaire study. Pregnancy Hypertens. 2016 Oct;6(4):350-355. doi: 10.1016/j.preghy.2016.08.232. Epub 2016 Aug 6. PMID 27939481
- [Background] Wright D, Poon LC, Rolnik DL, Syngelaki A, Delgado JL, Vojtassakova D, de Alvarado M, Kapeti E, Rehal A, Pazos A, Carbone IF, Dutemeyer V, Plasencia W, Papantoniou N, Nicolaides KH. Aspirin for Evidence-Based Preeclampsia Prevention trial: influence of compliance on beneficial effect of aspirin in prevention of preterm preeclampsia. Am J Obstet Gynecol. 2017 Dec;217(6):685.e1-685.e5. doi: 10.1016/j.ajog.2017.08.110. Epub 2017 Sep 6. PMID 28888591
- [Background] Shanmugalingam R, Hennessy A, Makris A. Aspirin in the prevention of preeclampsia: the conundrum of how, who and when. J Hum Hypertens. 2019 Jan;33(1):1-9. doi: 10.1038/s41371-018-0113-7. Epub 2018 Sep 19. PMID 30232399
- [Background] Ngo TTM, Moufarrej MN, Rasmussen MH, Camunas-Soler J, Pan W, Okamoto J, Neff NF, Liu K, Wong RJ, Downes K, Tibshirani R, Shaw GM, Skotte L, Stevenson DK, Biggio JR, Elovitz MA, Melbye M, Quake SR. Noninvasive blood tests for fetal development predict gestational age and preterm delivery. Science. 2018 Jun 8;360(6393):1133-1136. doi: 10.1126/science.aar3819. PMID 29880692
- [Background] Koh W, Pan W, Gawad C, Fan HC, Kerchner GA, Wyss-Coray T, Blumenfeld YJ, El-Sayed YY, Quake SR. Noninvasive in vivo monitoring of tissue-specific global gene expression in humans. Proc Natl Acad Sci U S A. 2014 May 20;111(20):7361-6. doi: 10.1073/pnas.1405528111. Epub 2014 May 5. PMID 24799715
- [Background] Roberge S, Nicolaides K, Demers S, Hyett J, Chaillet N, Bujold E. The role of aspirin dose on the prevention of preeclampsia and fetal growth restriction: systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Feb;216(2):110-120.e6. doi: 10.1016/j.ajog.2016.09.076. Epub 2016 Sep 15. PMID 27640943
- [Background] Seidler AL, Askie L, Ray JG. Optimal aspirin dosing for preeclampsia prevention. Am J Obstet Gynecol. 2018 Jul;219(1):117-118. doi: 10.1016/j.ajog.2018.03.018. Epub 2018 Mar 26. No abstract available. PMID 29588190
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Perneby C, Vahter M, Akesson A, Bremme K, Hjemdahl P. Thromboxane metabolite excretion during pregnancy--influence of preeclampsia and aspirin treatment. Thromb Res. 2011 Jun;127(6):605-6. doi: 10.1016/j.thromres.2011.01.005. Epub 2011 Feb 12. No abstract available. PMID 21316743
- [Background] Vainio M, Riutta A, Koivisto AM, Maenpaa J. Prostacyclin, thromboxane A and the effect of low-dose ASA in pregnancies at high risk for hypertensive disorders. Acta Obstet Gynecol Scand. 2004 Dec;83(12):1119-23. doi: 10.1111/j.0001-6349.2004.00396.x. PMID 15548142
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 203: Chronic Hypertension in Pregnancy. Obstet Gynecol. 2019 Jan;133(1):e26-e50. doi: 10.1097/AOG.0000000000003020. PMID 30575676
- [Background] Perni U, Sison C, Sharma V, Helseth G, Hawfield A, Suthanthiran M, August P. Angiogenic factors in superimposed preeclampsia: a longitudinal study of women with chronic hypertension during pregnancy. Hypertension. 2012 Mar;59(3):740-6. doi: 10.1161/HYPERTENSIONAHA.111.181735. Epub 2012 Feb 6. PMID 22311907
- [Derived] Khander A, Thomas C, Matthews K, Christos P, Alcus C, Alam T, Bush L, Deshmukh D, Chasen ST, Riley LE, Skupski DW, August P, Malha L. Comparison of 162 mg and 81 mg Aspirin for Prevention of Preeclampsia: A Randomized Controlled Trial. Obstet Gynecol. 2026 Jan 1;147(1):87-96. doi: 10.1097/AOG.0000000000006100. Epub 2025 Oct 24. PMID 41296512
- [Derived] Khander A, Matthews K, Christos P, Thomas C, Alam T, Alcus C, Bush L, Edusei E, August P, Malha L. Randomised controlled trial comparing low doses of aspirin in the prevention of pre-eclampsia (ASAPP): a study protocol. BMJ Open. 2025 Jul 8;15(7):e096779. doi: 10.1136/bmjopen-2024-096779. PMID 40633954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 81mg ASA | 162mg ASA
Started | 200 | 200
Completed | 181 (with pregnancy proceeding beyond 20 weeks and with delivery data available) | 184 (with pregnancy proceeding beyond 20 weeks and with delivery data available)
Not Completed | 19 | 16

BASELINE CHARACTERISTICS:
Population: All randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | 81mg ASA | 162mg ASA | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [32 to 38] | 35 [32 to 37] | 35 [32 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 200 | 400
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 46 | 78
  Not Hispanic or Latino | 150 | 140 | 290
  Unknown or Not Reported | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 41 | 31 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 38 | 81
  White | 61 | 77 | 138
  More than one race | 26 | 39 | 65
  Unknown or Not Reported | 27 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Preterm (<37 Weeks) Preeclampsia
Description: The incidence of preterm (<37 weeks) preeclampsia in high risk pregnant women treated with either 81 mg or 162 mg of daily aspirin during pregnancy.
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Population: Intention to treat analysis of all participants with pregnancy progressing beyond 20 weeks with delivery data available
Measure: Count of Participants; unit: Participants
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
Participants | 22 | 16
Statistical Analysis 1: Comparison: 81mg ASA vs 162mg ASA; Test type: Superiority; p = 0.28, Chi-squared; Risk Difference (RD) = 0.035 — Risk difference direction = 81mg arm minus 162mg arm

2. Primary Outcome: Incidence of Preeclampsia With Severe Features
Description: The incidence of preeclampsia with severe features (American College of Obstetricians and Gynecologists 2019 definition) in high-risk pregnant women treated with either 81 mg or 162 mg of daily aspirin during pregnancy.
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Population: Intention to treat analysis of all participants with pregnancy progressing beyond 20 weeks with delivery data available
Measure: Count of Participants; unit: Participants
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
Participants | 26 | 20
Statistical Analysis 1: Comparison: 81mg ASA vs 162mg ASA; Test type: Superiority; p = 0.31, Chi-squared; Risk Difference (RD) = 0.035 — Risk difference direction = 81mg arm minus 162mg arm

3. Primary Outcome: Composite Primary Outcome
Description: Composite of preterm preeclampsia and/or preeclampsia with severe features
Time Frame: 9 months for each participant
Population: Intention to treat analysis of all participants with pregnancy progressing beyond 20 weeks with delivery data available
Measure: Count of Participants; unit: Participants
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
Participants | 28 | 25
Statistical Analysis 1: Comparison: 81mg ASA vs 162mg ASA; Test type: Superiority; p = 0.61, Chi-squared; Risk Difference (RD) = 0.019 — Risk difference direction = 81mg arm minus 162mg arm

4. Secondary Outcome: Aspirin Adherence
Description: Evaluate and compare the adherence of pregnant women to 81mg and 162mg of daily low-dose aspirin using a validated, Simplified Medication Adherence Questionnaire (SMAQ).
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Population: Intention to treat analysis of all participants with pregnancy progressing beyond 20 weeks with delivery data available for adjudication and with SMAQ data available
Measure: Count of Participants; unit: Participants
Groups:
- 81mg ASA: Participants on 81mg of Aspirin a day
- 162mg ASA: Participants on 162mg of Aspirin a day
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
Participants
  20 weeks | 106 | 122
  26 weeks: number analyzed (Participants) | 136 | 139
  26 weeks | 124 | 126
  36 weeks: number analyzed (Participants) | 115 | 110
  36 weeks | 107 | 101

5. Secondary Outcome: Maternal and Fetal Outcomes
Description: Compare maternal and fetal outcomes in pregnant women at a high risk for preeclampsia who are treated with either 81mg or 162mg of daily aspirin during pregnancy, including gestational hypertension, postpartum hypertension, preterm delivery <37 weeks, fetal growth restriction (IUGR) or low birthweight (<2000g), placental abruption, ICU admission (maternal and neonatal), and maternal/fetal mortality.
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Population: Intention to treat analysis of all participants with pregnancy progressing beyond 20 weeks with delivery data available
Measure: Count of Participants; unit: Participants
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
Participants
  gestational Hypertension | 36 | 36
  maternal ICU admission | 2 | 1
  NICU admissions | 27 | 33
  postpartum Hypertension | 23 | 22
  Placental abruption | 0 | 8
  preterm delivery (<37 week) | 50 | 57
  IUGR or low birthweight | 21 | 16

6. Secondary Outcome: Time-to-event for Preeclampsia: Gestational Age at Onset of Preeclampsia
Description: Compare the time-to-event for developing preeclampsia for women treated with 81mg vs 162mg of aspirin per day. The time to event analysis will be made using the gestational age at the onset of preeclampsia as a variable
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Population: Intention to treat analysis of all participants with pregnancy progressing beyond 20 weeks with delivery data available
Measure: Mean (Standard Deviation); unit: weeks to developing preeclampsia
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
weeks to developing preeclampsia | 34.1 (5.08) | 34.3 (5.59)
Statistical Analysis 1: Comparison: 81mg ASA vs 162mg ASA; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = -0.20

7. Secondary Outcome: Aspirin Adherence- All Time Points Together
Description: To assess the adherence to low dose aspirin in pregnant women that are at high risk for preeclampsia and compare compliance rates for women on 81mg vs 162mg of aspirin per day using urine studies for salicylates and serum analysis. All time points together
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Population: All available SMAQ adherence questionnaires are considered from all timepoints cumulatively
Measure: Number; unit: surveys reporting adherence
Units Other Than Participants: Surveys
Arm/Group | 81mg ASA | 162mg ASA
Number analyzed (Participants) | 181 | 184
Number analyzed (Surveys) | 369 | 387
surveys reporting adherence | 337 | 349

8. Other Pre Specified Outcome: Impact of Co-morbidities on Incidence of Preeclampsia
Description: Assess the impact of specific co-morbidities (diabetes, chronic hypertension, renal disease and autoimmune disease), blood pressure control, age and race on the relationship between treatment group (81mg vs 162mg aspirin per day) and preeclampsia incidence.
Time Frame: 9 months for each patient (from recruitment until 6 weeks postpartum)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | 81mg ASA | 162mg ASA
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/184
Serious Adverse Events (participants affected / at risk) | 2/181 | 4/184
Other Adverse Events (participants affected / at risk) | 55/181 | 109/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 81mg ASA (N=181) | 162mg ASA (N=184)
Antepartum Fetal demise after 20 weeks (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) — Fetal demise reported after 20 weeks
Perinatal demise (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Perinatal demise due to congenital cardiomyopathy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 81mg ASA (N=181) | 162mg ASA (N=184)
Hypertension (Cardiac disorders) | 29 (29) | 47 (47) — Participant presented for unscheduled visit because of elevated blood pressure during the study period
Fetal concerns (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 19 (19) — Participant sent to triage for concerns about fetal movement or Non-stress test tracings
Vaginal Spotting (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 18 (18) — Participant with unscheduled visit because of vaginal bloody discharge or spotting
COVID (Infections and infestations) | 4 (4) | 14 (14) — Participant with unscheduled visit for documented COVID infection
Infection (Infections and infestations) | 7 (7) | 11 (11) — Participant with unscheduled visit because of concern for infection either viral or bacterial, non-COVID related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT04070573/Prot_SAP_000.pdf